CLINICAL TRIAL: NCT06672146
Title: A Randomized Phase II Trial of ASTX727 and Venetoclax Compared With ASTX727, Venetoclax, and Enasidenib for Newly Diagnosed Older Adults With IDH2 Mutant Acute Myeloid Leukemia: A MyeloMATCH Substudy
Brief Title: Comparing New Treatments for People With Newly Diagnosed Acute Myeloid Leukemia That Has an IDH2 Gene Change (A MyeloMATCH Treatment Trial)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - Safety Run-In Analysis
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-08951; NCI-2024-08951 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MM1OA-S03 (Other: SWOG); MM1OA-S03 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; decitabine and cedazuridine drug combination; enasidenib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (ASTX727 + venetoclax) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow aspiration, and bone marrow biopsy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax
- Arm 2 (ASTX727 + venetoclax + enasidenib) (Experimental): Patients receive ASTX727 PO QD on days 1-5, venetoclax PO QD on days 1-28, and enasidenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow aspiration, and bone marrow biopsy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Enasidenib; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
Drug: Enasidenib — Given PO
  Other Names: AG 221; AG-221; AG221; CC-90007 Free Base
  Arms: Arm 2 (ASTX727 + venetoclax + enasidenib)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II MyeloMATCH treatment trial studies how well ASTX727 and venetoclax plus enasidenib works compared to ASTX727 and venetoclax alone for the treatment of older patients with newly diagnosed acute myeloid leukemia (AML) or younger patients who are considered unfit for standard treatment, and who have an abnormal change (mutation) in the IDH2 gene. This gene mutation can cause AML to grow and spread. This trial is being done to see if adding enasidenib to the usual treatment can help more patients with the IDH2 gene get rid of AML.

ASTX727 is a fixed-dose formulation of two drugs, cedazuridine and decitabine. Cedazuridine is in a class of medications called cytidine deaminase inhibitors. It prevents the breakdown of decitabine, making it more available in the body so that decitabine will have a greater effect. Decitabine is in a class of medications called hypomethylation agents. It works by helping the bone marrow produce normal blood cells and by killing abnormal cells in the bone marrow. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Enasidenib works by stopping the growth and spread of tumor cells that have the IDH2 mutation. Giving ASTX727 and venetoclax plus enasidenib may work better in treating AML patients with the IDH2 mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of decitabine and cedazuridine (ASTX727) + venetoclax + enasidenib (Arm 2) before initiating randomization.

II. To compare the rate of measurable residual disease (MRD) negative complete remission (CR) based on multiparameter flow cytometry (MFC) after two cycles of treatment in older adults (or unfit adults age 18 or older) with IDH2 mutated Acute Myeloid Leukemia (AML) who receive ASTX727, venetoclax, and enasidenib versus ASTX727 and venetoclax alone.

SECONDARY OBJECTIVES:

I. To estimate the composite remission rate (CR + complete remission with incomplete count recovery [CRi] + complete remission with partial hematologic recovery [CRh]), relapse-free survival (RFS), event-free survival (EFS), duration of response (DOR), and overall survival (OS) of participants by treatment arm.

II. To estimate IDH2 mutated variant allele frequency, flow cytometry MRD, and molecular MRD after two cycles of therapy in participants' bone marrow aspirates and blood by treatment arm.

III. To estimate remission rates (CR with and without MRD [MFC and molecular MRD], CRh and CRi), and to estimate the rates of hematologic improvement by treatment arm.

IV. To estimate the frequency and severity of adverse events by treatment arm. V. To evaluate the association between MFC and molecular MRD after two cycles of protocol treatment with the outcomes RFS and OS (landmarked by date of MRD measurement) by treatment arm.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive ASTX727 orally (PO) once daily (QD) on days 1-5 and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive ASTX727 PO QD on days 1-5, venetoclax PO QD on days 1-28, and enasidenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

All patients undergo blood sample collection, bone marrow aspiration, and bone marrow biopsy throughout the trial.

After completion of study treatment, patients are followed up every month for the first year, every 2 months for the second year, every 3 months for the third year, and every 6 months until 5 years after registration or death.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been registered to the MYELOMATCH Master Screening and Reassessment Protocol prior to consenting to this study. Participants must have disease with a detectable IDH2 mutation based on central testing through the MYELOMATCH and be assigned to this clinical trial via MATCHBox prior to registration to this study

  * Note: Pre-enrollment/diagnosis labs must have already been performed under MYELOMATCH
* Participants must have newly diagnosed, untreated acute myeloid leukemia (AML) defined by having ≥ 20% blasts in the bone marrow and/or peripheral blood, excluding acute promyelocytic leukemia (APL) with PML-RARA
* Participants must not be receiving or planning to receive any other investigational agents while on protocol therapy
* Participants must not have received prior therapy for AML or myelodysplastic syndrome (MDS) and/or myeloproliferative neoplasm (MPN) with the exception of hydroxyurea, all-trans retinoic acid (ATRA), colony-stimulating factors, erythropoiesis-stimulating agents, immunosuppressive therapy, intrathecal chemotherapy, a single dose of cytarabine for cytoreduction, and/or leukapheresis
* Participants must not be currently receiving any cytarabine-containing therapy other than up to 1 g/m^2 of cytarabine, which is allowed for urgent cytoreduction. The use of prior hydroxyurea, all-trans retinoic acid (ATRA), BCR-ABL directed tyrosine kinase inhibitor, erythropoiesis-stimulating agent, thrombopoietin receptor agonist and lenalidomide are allowed. Participants may receive hydroxyurea prior to treatment assignment on this substudy for cytoreduction but must agree to discontinue hydroxyurea prior to beginning treatment on this substudy

  * White blood cell (WBC) must be < 25 x 10^9/L. Hydroxyurea, leukapheresis, and cytarabine < 1 g/m^2 are permitted to control the WBC prior to enrollment and initiation of protocol-defined therapy but must be stopped prior to initiation of protocol therapy
* Participants must be ≥ 60 years old; OR must be ≥ 18 years old and considered not eligible for cytarabine-based induction therapy
* Participants must have Zubrod Performance Status of 0-3 as determined by a history and physical (H&P) exam completed within 14 days prior to registration
* Participants must have a complete medical history and physical exam within 14 days prior to registration
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) unless history of Gilbert's syndrome. Participants with history of Gilbert's syndrome must have total bilirubin ≤ 3 x institutional ULN (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN, unless considered to be elevated due to disease involvement (within 14 days prior to registration)
* Participants must have adequate kidney function as evidenced by creatinine clearance ≥ 30mL/min (by Cockcroft Gault) within 14 days prior to registration
* Participants must not have a baseline corrected QT interval ≥ 480 msec using Fridericia correction (QTcF).

  * NOTE: Since older participants are at risk for prolonged QTc and may require supportive care with agents that affect QTc, an electrocardiogram (ECG) is recommended if clinically indicated. If the QTc is prolonged, they should be treated on MYELOMATCH TAP instead of MM1OA-S03
* Participants must have adequate cardiac function in the assessment of their treating physician. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2 or better
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to registration
* Participants with a known history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to registration, if indicated
* Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to registration, if indicated
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must be able to swallow and retain oral medications and have no known gastrointestinal disorders likely to interfere with absorption of oral medications
* Participants must have agreed to have specimens submitted for translational medicine for MRD under MYELOMATCH and specimens must be submitted

  * Enrollment to this treatment study requires prior enrollment into the myeloMATCH Master Protocol (MYELOMATCH). Participants enrolled in MYELOMATCH will submit bone marrow samples, peripheral blood samples, and buccal swabs to the Molecular Diagnostics Network (MDNet), the Clinical Laboratory Improvement Act (CLIA) laboratory network for myeloMATCH
  * In addition to the MYELOMATCH specimens, there will be specimens obtained on treatment for this substudy. These specimens will be derived from procedures performed as part of standard assessments in the clinical care and management of AML with material being sent to the MDNet laboratories as specified. After performing the required tests on the specimens, the MDNet laboratories will send the residual material for biobanking and future research. Therefore, participants must be asked for their consent for the biobanking of specimens for future unspecified research. Participants may refuse this, but it is mandatory for sites to ask participants
* Participants must be offered the opportunity to participate in specimen banking
* NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease negative (MRDneg) complete remission (CR) rate | Baseline to 5 years
  A randomized design will be used to compare binary endpoints in two arms with a single interim futility analysis. For the final analysis, a 2-sample proportion z-test will be used to compare the MRDneg-CR rates between arms with a two-sided alpha of 20%.

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | Baseline to 5 years
  Survival endpoints will be estimated using the Kaplan-Meier method and compared between arms using the log-rank test. Landmark survival endpoints after 2- and 4-cycles of therapy will be estimated using the Kaplan-Meier method. Time-dependent Cox regression models with response as a time-dependent covariate will be fit. Landmark Kaplan-Meier plots will be used describe marker associations with overall survival (OS) and RFS. Landmark and time-dependent Cox regression models will be fit with marker values as covariates. If endpoints subject to competing risks are analyzed, non-parametric cumulative incidence rates will be calculated, and associations will be evaluated using cause-specific hazard models
Event-free survival | Baseline to 5 years
  Survival endpoints will be estimated using the Kaplan-Meier method and compared between arms using the log-rank test. Landmark survival endpoints after 2- and 4-cycles of therapy will be estimated using the Kaplan-Meier method. Time-dependent Cox regression models with response as a time-dependent covariate will be fit. Molecular and flow MRD rates in the peripheral blood will be tabulated and summarized by arm. Landmark and time-dependent Cox regression models will be fit with marker values as covariates. If endpoints subject to competing risks are analyzed, non-parametric cumulative incidence rates will be calculated, and associations will be evaluated using cause-specific hazard models
Duration of response | Baseline to 5 years
  Response and toxicity rates will be tabulated. Survival endpoints will be estimated using the Kaplan-Meier method and compared between arms using the log-rank test. Landmark survival endpoints after 2- and 4-cycles of therapy will be estimated using the Kaplan-Meier method. Time-dependent Cox regression models with response as a time-dependent covariate will be fit. Landmark and time-dependent Cox regression models will be fit with marker values as covariates. If endpoints subject to competing risks are analyzed, non-parametric cumulative incidence rates will be calculated, and associations will be evaluated using cause-specific hazard models
OS | Baseline to 5 years
  Survival endpoints will be estimated using the Kaplan-Meier method and compared between arms using the log-rank test. Landmark survival endpoints after 2- and 4-cycles of therapy will be estimated using the Kaplan-Meier method. Time-dependent Cox regression models with response as a time-dependent covariate will be fit. Molecular and flow MRD rates in the peripheral blood will be tabulated and summarized by arm. Landmark Kaplan-Meier plots will be used describe marker associations with OS and RFS. Landmark and time-dependent Cox regression models will be fit with marker values as covariates. If endpoints subject to competing risks are analyzed, non-parametric cumulative incidence rates will be calculated, and associations will be evaluated using cause-specific hazard models

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Huselton, Principal Investigator — SWOG Cancer Research Network
Locations (86):
- United States (84):
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills Health Center, San Mateo, California
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - MaineHealth Cancer Care and IV Therapy - Brunswick, Brunswick, Maine
  - Mid Coast Hospital, Brunswick, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm